CLINICAL TRIAL: NCT03023358
Title: Compared the Efficacy and Safety of CDOP Combined With Chidamide and CDOP in de Novo Peripheral T Cell Lymphoma Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Ru Feng, Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDOP201602
Record Dates: First submitted 2016-11-03; First posted 2017-01-18 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Peripheral T Cell Lymphoma
Keywords: peripheral T cell lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Cyclophosphamide; liposomal doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- chidamide regimen (Experimental): patients receive chidamide (30mg twice every week) po, cyclophosphamide (750mg/m2) iv on day 1, liposomal doxorubicin (30mg/m2) iv on day 1, vincristine (1.4mg/m2, max to 2mg) iv on day 1 and prednisone (100mg/d) po on day 1-5.
  Interventions: Drug: chidamide; Drug: cyclophosphamide; Drug: liposomal doxorubicin; Drug: vincristine; Drug: prednisone
- CDOP regimen (Active Comparator): patients receive cyclophosphamide (750mg/m2) iv on day 1, liposomal doxorubicin (30mg/m2) iv on day 1, vincristine (1.4mg/m2, max to 2mg) iv on day 1 and prednisone (100mg/d) po on day 1-5.
  Interventions: Drug: cyclophosphamide; Drug: liposomal doxorubicin; Drug: vincristine; Drug: prednisone

INTERVENTIONS:
Drug: chidamide — 30mg po twice a week
  Other Names: epidaza
  Arms: chidamide regimen
Drug: cyclophosphamide — 750mg/m2 iv on day 1
Drug: liposomal doxorubicin — 30mg/m2 iv on day 1
Drug: vincristine — 1.4mg/m2 iv on day 1
Drug: prednisone — 100mg/d po on day 1-5

SUMMARY:
The prognosis for Peripheral T cell lymphomas (PTCL) remains poor in comparison to B cell NHL. This is largely due to lower response rates and less durable responses to standard combination chemotherapy regimens such as CHOP. Whether CDOP plus Chidamide can improve the prognosis for PTCL.

DETAILED DESCRIPTION:
Peripheral T-cell lymphomas (PTCL) are a heterogeneous group of lymphoproliferative disorder arising from mature T-cells of post-thymic origin. PTCL represent a relatively uncommon group of hematologic malignancies within non-Hodgkin lymphomas (NHL), accounting for about 10% of NHL cases. The prognosis for PTCL remains poor in comparison to B-cell NHL. This is largely due to lower response rates and less durable responses to standard combination chemotherapy regimens such as CHOP. Progress has been further hampered by the relative rarity and the biological heterogeneity of the diseases. Among PTCL cases worldwide, the most common subtypes include PTCL-not otherwise specified (PTCL-NOS; 26%), angioimmunoblastic T-cell lymphoma (AITL; 18.5%), NK/T-cell lymphoma (10%), adult T-cell leukemia/lymphoma (ATLL; 10%), ALK-positive anaplastic large cell lymphoma (ALCL; 7%) and ALK-negative ALCL (6%); subtypes such as enteropathy-associated T-cell lymphoma (EATL; <5%) and primary cutaneous ALCL are relatively rare (<2%) with ALCL more common than NK/T or ATLL in the United States.

PTCLs are less responsive to and have less frequent durable remissions with standard chemotherapy regimens such as CHOP and thus carry a poorer prognosis compared to diffuse large B-cell lymphomas. In prospective randomized studies, PTCLs have been included with aggressive B-cell lymphomas. However, it has not been possible to assess the impact of chemotherapy in this subgroup of patients with PTCLs due to small sample size. Only limited data exist from randomized trials comparing the efficacy of chemotherapy regimens exclusively in patients with PTCL.

CHOP chemotherapy is the most commonly used first-line regimen for patients with PTCL. However, with the exception of ALK+ ALCL, outcomes are disappointing compared to the favorable results achieved with DLBCL. Chemotherapy regimens that are more intensive than CHOP have not shown any significant improvement in OS in patients with PTCL, with the exception of ALCL.

CHOP chemotherapy is frequently curative in only the small number of patients with favorable prognostic features. As previously discussed, retrospective analysis from the International T-cell Lymphoma Project showed that anthracycline-based chemotherapy did not favorably impact survival in patients with the most common forms of PTCLs, namely PTCL-NOS and AITL. In a retrospective study conducted by the British Columbia cancer agency, the 5-year OS rate for patients with PTCL-NOS primarily treated with CHOP or CHOP-like regimens was only 35%; among these patients, the 5-year OS rates were higher in patients with low-risk IPI scores compared with those with high-risk IPI scores (64% vs. 22%, respectively). In addition, patients with ALK-positive ALCL had superior clinical outcome compared to those with ALK-negative ALCL (5-year OS 58% vs. 34%, respectively). The addition of etoposide to CHOP (CHOEP regimen) compared with CHOP alone was evaluated in a randomized study by the German High-grade NHL Study Group (DSHNHL). In relatively young patients with favorable prognosis aggressive NHL (age ≤60 years; normal LDH levels), the CHOEP regimen resulted in significantly higher CR rate (88% vs. 79%; P=0.003) and 5-year EFS rate (69% vs. 58%; P=0.004). No difference was observed in OS outcomes between the regimens. It should also be noted that in this study, the majority of patients had B-cell histology, with only 14% diagnosed with T-cell NHL (with 12% of patients having ALCL, PTCL-NOS, or AITL histology).36 In an analysis of a large cohort of patients with PTCL treated within the DSHNHL trials, patients with ALK- positive ALCL had favorable outcomes with CHOP or CHOP with etoposide (CHOEP). Three-year EFS and OS rates were 76% and 90%, respectively, for patients with ALK-positive ALCL. The corresponding outcomes were 50% and 67.5%, respectively, for AITL, 46% and 62%, respectively, for ALK-negative ALCL and 41% and 54%, respectively, for PTCL-NOS. Among those with T-cell lymphoma, CHOEP was associated with a trend for improved EFS among relatively young patients (age <60 years) and is an option for these patients. CHOP-21 appeared to be the standard regimen for patients age >60 years, given that the addition of etoposide did not provide an advantage in these older patients due to increased toxicity. Among patients with ALK-negative ALCL, AITL and PTCL-NOS, those with low-risk IPI scores (IPI <1) had a relatively favorable prognosis; contrastingly, patients with higher risk IPI scores derived minimal benefit from CHOP or CHOEP.

Histone deacetylases (HDACs) are involved in the remodeling of chromatin and play a key role in the epigenetic regulation of gene expression. HDACs act as transcription repressors by removing acetyl groups from the e-amino- terminus of lysine residues within histones to promote tighter winding of DNA around histone proteins. Elevated expression or activity of HDACs is implicated in the development and progression of cancer. Inhibition of HDAC enzymes results in increased histone acetylation, thereby inducing an open chromatin conformation and transcription of previously dormant genes. At least 18 human HDACs have been identified and are grouped into four classes. HDAC enzymes class I (HDAC1, 2, 3, and 8), class II (HDAC4, 5, 7, and 9 as IIa, and HDAC6 and 10 as IIb), and class IV (HDAC11) utilize a zinc-catalyzed mechanism for deacetylation of histones and non-histone proteins, whereas class III (SIRT 1-7) HDACs are NAD+ dependent deacetylase enzymes. Although the precise biological functions of individual HDACs are still largely unknown, the importance of HDAC enzymes in the malignant phenotype has been most closely associated with Class I HDACs 1-3. In addition, Class IIb HDACs 6 and 10 have been found to play a role in the expression and stability of tumor angiogenesis gene products.

The synthesis of small-molecule HDAC inhibitors (HDACi) has been an active focus in the field of anticancer drug discovery in recent years. Several different chemical classes of HDACi have been described, including hydroxamic acids, carboxylic or short-chain fatty acids, cyclic peptides, and benzamides. Examples of each of these classes have entered clinical development as antitumor agents. Among them, the hydroxamic acid vorinostat (SAHA) and cyclic peptide romidepsin (FK-228) were approved in the United States for the treatment of cutaneous T-cell lymphoma, and very recently, romidepsin for peripheral T-cell lymphoma.

chidamide (CS055/HBI-8000), a new member of the benzamide class of HDACi. Chidamide inhibits HDAC1, 2, 3, and 10 in the low nanomolar concentration range with broad spectrum antitumor activity in vitro and in vivo. Mechanism studies have demonstrated that chidamide stimulates human immune cell-mediated tumor cell killing activity with increased expression of genes and proteins involved in natural killer (NK) cell functions.

Chidamide was found to be a low nanomolar inhibitor of HDAC1, 2, 3, and 10, the HDAC isotypes well documented to be associated with the malignant phenotype. Significant and broad spectrum in vitro and in vivo anti- tumor activity, including a wide therapeutic index, was observed. Chidamide was also shown to enhance the cytotoxic effect of human peripheral mononuclear cells ex vivo on K562 target cells, accompanied by the upregulation of proteins involved in NK cell functions. Furthermore, the expression of a number of genes involved in immune cell- mediated antitumor activity was observed to be upregulated in peripheral white blood cells from two T-cell lymphoma patients who responded to chidamide administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years are eligible.
* Patients must be diagnosed of de love peripheral T cell lymphoma (include PTCL not otherwise specified, angioimmunoblastic T cell lymphoma, ALK negative anapestic large cell lymphoma and enteropathy-associated T cell lymphoma). Patients must be chemo-naive.
* ECOG PS of 0, 1, 2 at screening.
* Serum biochemical values with the following limit: - creatine </= 2.0 mg/dl, - total bilirubin </= 2.0mg/dl, - transaminases (SG PT) </= 3X ULN
* Ability to understand an provide signed informed consent.

Exclusion Criteria:

* Presence of active systemic infection.
* Any coexisting medical condition that in the judgment of the treating physician is likely to interfere with study procedures or results.
* Nursing women, women of childbearing potential with positive urine pregnancy test, or women of childbearing potential who are not willing to maintain adequate contraception (such as birth control pills, IUD, diaphragm, abstinence, or condoms by their partner) over the entire course of the study.
* Patients whom the investigators considered were not applicable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2017-02; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
complete remission rate | 3 year

SECONDARY OUTCOMES:
disease free survival | 3 years
overall survival | 3 years
time to progression | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ru Feng, M.D., Study Chair — Department of Hematology Nanfang Hospital, The Southern Medical University
Locations (1):
- Ru Feng, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shi Y, Dong M, Hong X, Zhang W, Feng J, Zhu J, Yu L, Ke X, Huang H, Shen Z, Fan Y, Li W, Zhao X, Qi J, Huang H, Zhou D, Ning Z, Lu X. Results from a multicenter, open-label, pivotal phase II study of chidamide in relapsed or refractory peripheral T-cell lymphoma. Ann Oncol. 2015 Aug;26(8):1766-71. doi: 10.1093/annonc/mdv237. Epub 2015 Jun 23. PMID 26105599
- See also: Nan fang Hospital, the Southern Medical University — http://www.nfyy.com/